CLINICAL TRIAL: NCT01834339
Title: A Randomized, Parallel-Group (Autogenous EVPOME Versus AlloDerm Without Incorporation of Keratinocytes) Study in Subjects Reconstructed With Large Defect Mandibular Resection in Need of Vestibuloplasty for Dental Rehabilitation
Brief Title: EVPOME Versus AlloDerm in Subjects Reconstructed With Large Defect Mandibular Resection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of cGMP facility to manufacture product used in clinical trial.
Sponsor: Stephen E. Feinberg (Other)
Responsible Party: Sponsor-Investigator, Stephen E. Feinberg, Professor & Associate Chair of Research, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00069761
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Mandibular Injuries
Keywords: vestibuloplasty
MeSH Terms: conditions — Mandibular Injuries | interventions — Alloderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AlloDerm (Active Comparator): The subject will be treated with the standard of care, AlloDerm, to cover the defect in the mouth.
  Interventions: Biological: AlloDerm
- EVPOME (Experimental): An ex-vivo produced oral mucose equivalent (EVPOME) will be used to cover the defect in the top of the mouth.
  Interventions: Biological: EVPOME

INTERVENTIONS:
Biological: AlloDerm
  Arms: AlloDerm
Biological: EVPOME
  Arms: EVPOME

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of performing oral reconstructive surgeries using either AlloDerm, a product commonly used for this purpose, or AlloDerm that has been overlaid with the subject's oral mucosal cells and developed into a type of graft that is called an ex vivo produced oral mucosal equivalent, EVPOME.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult over 18 years of age
* Have a free fibular graft placed more than six months ago that has been used for restoration of mandibular continuity.
* Be in need of surgery to increase the vestibular fold of the grafted mandible for placement of a dental prosthesis to restore function

Exclusion Criteria:

* Any liver, kidney, heart, blood, metabolic or systemic disease which may make execution of the protocol of interpretation of the results difficult
* A history of syphilis, HIV, Hepatitis B or Hepatitis C
* Pregnancy or planning to become pregnant
* Known or suspected allergy to bovine (cow) protein
* Receiving radiation
* Currently smoking or using tobacco products
* Talking medication that can result in gingival enlargement (Cyclosporine, Dilantin, calcium channel blockers)
* Allergy to any of the following antibiotics Gentamycin, Cefoxitin, Lincomycin, Polymyxin B, Vancomycin, cephalosporins, or clindamycin
* Allergy to Polysorbate 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent Graft Contracture | 2-24 weeks
  During surgery, after preparation of the recipient bed, the recipient bed and the graft will be measured for the maximum distance between non-resorbable sutures placed at the margins of the graft. Post-surgical measurements of the graft site will be taken at visits 5, 6, 7, and 8 and compared to original graft size to assess percentage of graft contracture.

SECONDARY OUTCOMES:
Degree of Epithelialized Tissue | 4 weeks after surgery
  Degree of epithelialized mucosa will be assessed by biopsy taken at the geometric center of the graft at week 4 s/p grafting. The biopsy will be evaluated by routine histology for the presence of an intact and stratified keratinized epithelial layer and by immunohistochemistry (IHC) for microvessel vascular ingrowth into the dermis/dermal matrix (AlloDerm).
Laser Doppler Flowmetry (LDF) | Visit 1 and 2 and 4 weeks after surgery
  LDF measurements will be used to assess graft blood flow (tissue perfusion of the grafts). The LDF measures will also be compared with the immunohistochemistry (IHC) results seen on the biopsy to determine the relationship between the flood flow and degree of microvessel infiltration into the dermis/dermal matrix (AlloDerm) based on the two measures.

OTHER OUTCOMES:
Graft Color | 4 weeks after surgery
  Graft color is correlated to vascular perfusion and thus can give us an indication of graft vascularity. Primarily we expect the color rendition to be similar to the surrounding tissue. Finger pressure will be applied in the center of the graft for 15 seconds and/or until tissue blanching. The pressure will then be released and the time for the tissue to return to its previous color will be timed. If the tissue returns to its previous color within 15 seconds, this will be recorded as positive graft vascularity. If not, then it will be recorded as negative graft vascularity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Feinberg, DDS, MS, PhD, Principal Investigator — Faculty
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No